CLINICAL TRIAL: NCT03991962
Title: Phase II Study to Evaluate Modified Folfirinox and Stereotactic Body Radiation Therapy in Non-metastatic Unresectable Pancreatic Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000024671
Record Dates: First submitted 2019-06-18; First posted 2019-06-19 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Open label, single group design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- mFOLFIRINOX followed by SBRT (Experimental): Patients will receive mFOLFIRINOX, followed stereotactic body radiotherapy (SBRT).
  Interventions: Drug: mFOLFIRINOX; Radiation: Stereotactic body radiotherapy (SBRT)

INTERVENTIONS:
Drug: mFOLFIRINOX — Patients will receive 6-12 cycles of mFOLFIRINOX every 2 weeks
Radiation: Stereotactic body radiotherapy (SBRT) — Stereotactic body radiotherapy (SBRT) will be delivered to the primary tumor and any adjacent involved lymph nodes to 33 Gy in 5 fractions over the course of 2 weeks, and within 4 weeks of chemotherapy.

SUMMARY:
The purpose of this study is to evaluate the efficacy of modified FOLFIRINOX followed by stereotactic body radiotherapy (SBRT) in patients with borderline resectable pancreatic cancer (BRPC) and locally advanced pancreatic cancer (LAPC). The primary hypothesis will be to determine if modified FOLFIRINOX followed by SBRT improves progression free survival (PFS) compared to historical controls treated with gemcitabine-based chemotherapy with or without standard fractionated radiation.

DETAILED DESCRIPTION:
The Primary and Secondary are listed below.

Primary Objective:

- To evaluate progression free survival after modified FOLFIRINOX and SBRT in borderline resectable and locally advanced pancreatic cancer.

Secondary Objective:

* To evaluate the radiographic response to FOLFIRINOX and SBRT by comparing IV contrast CT scans before and after therapy.
* To determine rates of recurrence (local only, systemic only, and both local and systemic), and overall survival.
* To determine rates of grade 3 or greater gastrointestinal toxicity, including acute toxicities occurring within 3 months of treatment, and late toxicities occurring over 3 months after completion of radiation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed pancreatic adenocarcinoma
* Borderline resectable pancreatic adenocarcinoma or locally advanced pancreatic adenocarcinoma
* No evidence of extrapancreatic disease on diagnostic imaging
* No evidence of invasion into the duodenum or stomach, as determined by EGD/EUS
* No prior treatment (chemotherapy, biological therapy, or radiotherapy) for pancreatic cancer
* No prior treatment with oxaliplatin, irinotecan, fluorouracil, or capecitabine
* ECOG Performance Status of 0-1
* No other malignancy within past five years (exceptions include basal cell carcinoma of the skin, cervical carcinoma in situ, and non-metastatic prostate cancer)
* No evidence of second malignancy at the time of study entry
* No interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* No > grade 2 sensory peripheral neuropathy
* No uncontrolled seizure disorder, active neurological disease, or known CNS disease
* No significant cardiac disease, including the following: unstable angina, New York Heart Association class II-IV congestive heart failure, myocardial infarction within six months prior to study enrollment
* Not pregnant and not nursing
* No other medical condition or reason that, in the opinion of the investigator, would preclude study participation
* Laboratory parameters as follows:

  * Absolute neutrophil count ≥1,500/uL,
  * Platelet count ≥75,000/uL,
  * Hemoglobin ≥9 g,/dL,
  * Creatinine <1.5 X ULN or estimated GFR >30 ml/min,
  * Bilirubin <1.5 X ULN,
  * AST and ALT <3 X ULN,
  * Negative pregnancy test in women of childbearing potential
* Able to be treated with SBRT only at the Smilow New Haven campus
* Able to have fiducials placed in the pancreas

Exclusion Criteria:

* Failing to meet any of the Inclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-09-24 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 9 months
  Progression-free survival (PFS) at will be judged by CT scan and Response evaluation criteria in solid tumors (RECIST).

SECONDARY OUTCOMES:
Radiographic Response | Within 21 days of starting study drug
  Radiographic response to FOLFIRINOX and SBRT will be done by comparing IV contrast CT scans before and after therapy.
Rates of Recurrence | Up to 3 years
  Rates of recurrence (local only, systemic only, and both local and systemic) will be monitored for up to 3 years depending on time when the initiation of treatment begins.
Rates of grade 3 or greater gastrointestinal toxicity | Up to 3 months post treatment
  Grade 3 or greater gastrointestinal toxicities will be monitored including acute toxicities occurring within 3 months of treatment, and late toxicities occurring over 3 months after completion of radiation.
Overall Survival | Up to 3 years
  Patients will be monitored for overall survival for up to 3 years depending on time when the initiation of treatment begins.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Johung, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No